CLINICAL TRIAL: NCT02380196
Title: The Utility of Circulating Tumor Cells as Confirmation of Pathologic Diagnosis in Patients With Suspected Early Stage Non-small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 02515
Record Dates: First submitted 2015-03-02; First posted 2015-03-05 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2019-07

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Collection
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary objective of this study is to determine whether circulating tumor cells (CTCs) can be used as a non-invasive means of confirming pathologic diagnosis in early-stage (Stage I) non-small cell lung cancer (NSCLC). Patients scheduled to undergo surgical intervention will have blood samples obtained to test for CTCs. Presence of CTCs will be compared to final pathologic diagnosis based on surgical specimens to assess the sensitivity of using CTCs alone to make a definitive diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of stage I NSCLC a. Only patients with a pathologically confirmed NSCLC will be retained for data analysis b. Should pathologic diagnosis reveal a more advanced stage, these subjects will remain in the study
2. 18 years of age
3. Ability to read and sign informed consent
4. Both men and women and members of all races and ethnic groups are eligible for this trial.

Exclusion Criteria:

1. Prior cancer diagnosis, excluding previously treated non-melanoma skin cancer
2. Prior or ongoing treatment of the clinically diagnosed cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-small cell lung cancer (NSCLC)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-03; Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Charles Simone, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States